CLINICAL TRIAL: NCT03935867
Title: New York University (NYU) Falls Prevention Program
Brief Title: New York University Falls Prevention Program
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Grant applications to fund the investigation were not selected for fundin4.
Sponsor: New York University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: S15-01199
Record Dates: First submitted 2019-04-30; First posted 2019-05-02 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2019-04

CONDITIONS: Falls Related Risk Factors in the Elderly

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- C-PROFET group (Experimental): Community-dwelling, older adults participating in a home-based program -- C-PROFET, our adaptation of Prevention Of Falls in the Elderly Trial (PROFET).
  Interventions: Behavioral: C-PROFET

INTERVENTIONS:
Behavioral: C-PROFET — An expansion of the evidence-based, multi-factorial, fall prevention program PROFET (Prevention Of Falls in the Elderly Trial), developed for older adults who experienced a fall-related injury, to an at risk community-dwelling population who have not sustained a fall-related injury requiring medical intervention.

SUMMARY:
Limited health services research and evidence-based programming has been focused on elderly fall prevention, despite high fall-related morbidity and mortality. Among NY's elderly population, falls account for nearly half of all older adults' injury-related deaths and are the 4th leading cause of hospitalizations. As fall risk increases with age, the magnitude of this health issue will continue to increase. Scientific evidence shows that prevention efforts significantly reduce the frequency and severity of falls. Research also suggests that multi-component intervention programs, such as Prevention Of Falls in the Elderly Trial, "PROFET", are successful because benefits are derived from small improvements across several risk categories.

The investigators propose expanding the reach of fall prevention efforts to at-risk and underserved populations of community-dwelling, older adults by delivering a home-based program -- "C-PROFET", an adaptation of Prevention Of Falls in the Elderly Trial (PROFET), an evidence-based, multi-factorial, fall prevention program. Investigators will test two hypotheses: (1) Oral health care programs and services can be a portal for identifying underserved community dwelling elders at risk for falls who can benefit from a fall prevention program; and (2) Provision of fall prevention efforts to an at-risk clinical population before these patients experience a serious fall-related injury will reduce fall-risk, and potentially decrease fall-related morbidity, mortality, and healthcare costs.

This initiative is to lay the necessary groundwork for larger implementation efforts that will advance efforts to reduce fall risk in vulnerable, community-dwelling older adults. The investigators propose to deliver "C-PROFET" to vulnerable, older adults identified through dental clinics and community oral health outreach services. The overall objectives are to improve patient-centered health outcomes, demonstrate feasibility of a multicomponent intervention to reduce/prevent fall-related morbidity and mortality in an at-risk, community-dwelling, clinical population, and disseminate this falls prevention program to community partner organizations to broadly translate these findings into clinical practice.

DETAILED DESCRIPTION:
Implementing innovative, cost-effective community-based delivery modalities that reliably and effectively deliver evidence-based, culturally-sensitive programs, proven to prevent injury, preserve function, improve quality of life, and reduce morbidity and mortality among an older and more diverse population, will significantly impact health costs and help address the anticipated surge in demand for health services and long-term care. Such efforts need to appeal to diverse populations and have outcomes achievable with a community delivery.

This application is proposing to expand the reach of an evidence-based program, "PROFET", developed for older adults who experienced a fall-related injury, to an at risk community-dwelling population who have not sustained a fall-related injury requiring medical intervention. The investigators hypothesize that oral health care programs and services can be a portal for identifying underserved community dwelling elders at risk for falls who can benefit from a fall prevention program. As more adults see their dentist than visit a physician in a given year, dental clinics, a safety net site for the delivery of oral health care to the elderly, are ideally situated to take an active role in injury prevention efforts. Dental clinics attached to community health centers and academic institutions have established linkages and referral patterns across systems of care and disciplines that can facilitate delivery of preventive services prior to an injury-sustaining event, delaying or preventing unintentional injuries. To date, fall prevention efforts have predominately targeted those who have already experienced an injury-sustaining fall. All older adults may profit from fall prevention interventions (regardless of whether they have experienced a fall-related serious injury). Expanding delivery to reach an at-risk population living in the community, will enable earlier intervention efforts to prevent/reduce falls, serious injury and hospital stays including a first serious fall which in and of itself increases risk for subsequent serious falls.

The aims of this initiative are to: (1) adapt and deliver "C-PROFET", an evidence-based, multifactor fall prevention program, to at-risk, community-dwelling older (65+), multi-ethnic, economically constrained, community residents (n=30) identified in non-traditional community settings (general dental clinic and community dental outreach program delivering oral health care to the elderly in community-based facilities, including senior centers); and (2) to assess the reach, uptake, feasibility and acceptability of the program. NYU College of Dentistry (NYUCD) dental clinic is a low cost community clinic providing quality dental care to the uninsured and those living on a restricted income. The clinic maintains over 300,000 patient visits annually and 17% of the patient population are 65 and older. Examination of the utility of the dental clinic and dental outreach program as a portal for fall prevention programs will be guided by the "RE-AIM" framework which consists of five core elements: (1) Reach ("How do investigators reach the targeted population?"); (2) Effectiveness ("How do investigators know the program is effective?); (3) Adoption ("How effective is this program in different settings?"); (4) Implementation ("How do investigators ensure that the program is delivered consistently?"); (5) Maintenance ("How do investigators incorporate the program so that it is delivered over the long term?").

ELIGIBILITY:
Inclusion Criteria:

1. Is 65 years of age or older
2. Lives in the New York metropolitan area
3. Lives in a private residence or assisted living apartment
4. Understands English
5. Has one or more fall risk factors
6. Has not had a prior fall-related injury requiring emergency care
7. Is cognitively competent and has the capacity to give consent

Exclusion Criteria:

1. Has had a prior fall related injury requiring emergency care
2. Will be unavailable for a home visit within the next 3 months

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07-29 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
A change in environmental falls-related risk factors in the home | 3 months
  A Home Hazards and Safety Assessment will be conducted to identify any fall-related hazards in the home by the C-PROFET. An Occupational Therapist will discuss with the subject the results and recommended changes to the home to minimize the risk of future falls. A brief follow-up telephone survey will be conducted within three months of the home visit to assess the participant's adherence and barriers to fall prevention recommendations and referral follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria H. Raveis, PhD, Principal Investigator — New York University
Locations (1):
- New York University College of Dentistry, New York, New York, United States

REFERENCES:
- [Background] Close J, Ellis M, Hooper R, Glucksman E, Jackson S, Swift C. Prevention of falls in the elderly trial (PROFET): a randomised controlled trial. Lancet. 1999 Jan 9;353(9147):93-7. doi: 10.1016/S0140-6736(98)06119-4. PMID 10023893
- [Background] Northridge ME, Nevitt MC, Kelsey JL, Link B. Home hazards and falls in the elderly: the role of health and functional status. Am J Public Health. 1995 Apr;85(4):509-15. doi: 10.2105/ajph.85.4.509. PMID 7702114